CLINICAL TRIAL: NCT04226534
Title: Constructing a Psychophysiological Database Towards the Optimization of the Methodological Approach During, and Training Advice After Maximal Effort Tests.
Brief Title: A Psychophysiological Database of Maximal Effort Tests.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Jo Ghillebert, Principle Investigator, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: VUB-BLITS
Record Dates: First submitted 2019-12-18; First posted 2020-01-13 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maximal effort test (Other): Physiological database
  Interventions: Other: Maximal effort test

INTERVENTIONS:
Other: Maximal effort test — Performing a maximal effort test on the treadmill

SUMMARY:
The aim of this study is first to construct a database containing psychophysiological data from athletes performing a maximal effort test. Second, the investigators want to use the data to optimize the methodological approach during, and trainings advice after maximal effort tests.

DETAILED DESCRIPTION:
The lab (and research group) of Human Physiology and Sports Physiotherapy of the Vrije Universiteit Brussel performs exercise tests in both trained and untrained populations. The aim of the maximal effort test is to evaluate endurance capacity and provide recommendations to monitor training load. Until now, this is done by objective parameters such as heart rate, speed, time, power, etcetera. Researchers already presented a method to quantify training intensity distribution in elite endurance athletes based on the rating of perceived exertion. However, during pilot testing and everyday experience, these cut-off values are not always applicable to each individual athlete, nor are they the same for different sports. Therefore, the investigators want to investigate the possible relation between the exercise intensity, and objective and subjective parameters. Thereafter, the investigators want to provide recommendations to a new way of methodological approach during, and trainings advice after maximal effort tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Trained
* No medication influencing heart rate or physical performance

Exclusion Criteria:

* Disease
* injury
* medication influencing (maximal) heart rate or exercise performance

Decision made after sports medical evaluation, comprising personal and family history, physical examination and resting electrocardiogram (ECG).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2040-01-01 (Estimated); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
Ergospirometry | Up to one hour
  oxygen consumption and carbon di-oxide production (ml/min/kg)

SECONDARY OUTCOMES:
blood samples | Up to one hour
  Lactate concentration (mmol)
Rating of perceived effort | Up to one hour
  Rating of Perceived exertion on a scale from six to twenty

CONTACTS AND LOCATIONS:
Overall Officials: Luk Buyse, Msc. dr., Principal Investigator — Vrije Universiteit Brussel, Human Physiology and Sports Physiotherapy
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided